CLINICAL TRIAL: NCT02205905
Title: An Open-label, Single-dose, Non-randomized Study of the Absorption, Metabolism, and Excretion of Intravenously Administered 14C-labeled PER977 in Healthy Male Subjects
Brief Title: An Open-label, Single-dose, Non-randomized Study of IV 14C-labeled PER977 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: World Wide Clinical Trials Early Phase Services, LLC (Unknown)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PER977-01-004
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2016-09

CONDITIONS: Healthy
Keywords: PER977; metabolic disposition; mass balance; metabolites; radiolabeled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 14C PER977 (Experimental): Open-label, single-dose, non-randomized study of 14C PER977 in six healthy male subjects
  Interventions: Drug: 14C PER977

INTERVENTIONS:
Drug: 14C PER977 — Open-label, single dose
  Other Names: ciraprantag

SUMMARY:
This is an open-label, single-dose, non-randomized study in healthy male subjects to characterize the mass balance, metabolic disposition, and identification of the metabolites and general metabolic pathways following administration of a single dose of IV solution containing 200 mg of PER977 plus a tracer amount of 14C PER977 in health male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. 18-55 years of age (inclusive)
3. Body mass index 18-32 kg/m2 (inclusive) and a minimum of 50 kg (110 lbs)
4. voluntarily consent to participate and provide written informed consent prior to start of study specific procedures
5. Willing and able to remain in the study unit for the entire duration of the confinement period
6. Willing to collect all urine and fecal samples for the duration of the study period as required
7. Will to eat entire meals and snacks provided during confinement at the research facility, and understand diet will include foods with high fiber content and possibly prune juice
8. Willing to use a waterless commode located in a designated dry room for urine and feces collection for the duration of the study period as required
9. Willing to abstain from showering for the first 72 hours following study drug administration. After the restriction is lifted, willing to provide a urine sample prior to showering for the remainder of the confinement period.

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any condition which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results
2. Clinically significant abnormal finding on the physical exam, medical history, electrocardiogram or clinical laboratory resutls at screening
3. History or presence of allergic or adverse response to anticoagulant reversal agents or related drugs
4. Significantly abnormal diet within 4 weeks
5. Donated blood or plasma within 30 days
6. Participated in another clinical trial (randomized subjects only) within 30 days
7. Participated in a radiolabeled clinical trial within the last 12 months
8. Used any over-the-counter medication, including nutritional supplements, within 7 days
9. Used any prescription medication within 14 days prior
10. Treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates,phenothiazines, cimetidine, carbamazepine, etc. within 30 days
11. Smoked or used tobacco products within 60 days
12. History of substance abuse or treatment (including alcohol ) within the past 2 years
13. Positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine at screening or check-in
14. Positive test for hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus at screening or has previously been treated for hepatitis B, hepatitis C or HIV infection
15. Has irregular bowel habits
16. Has had significant radiation exposure within the prior 12 months

Ages: 15 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mass balance of PER977 and metabolite | 3 weeks
  To characterize the mass balance, metbaolic disposition, and identification of the metabolites and general metabolic pathways following administration of a single dose of IV solution containing 200 mg of PER977 plus a tracer amount of 14C PER977 to healthy male subjects

SECONDARY OUTCOMES:
Number of subjects with adverse events | 3 weeks
  To assess the safety and tolerability of a single intravenous dose of 200 mg PER977

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Zamora, MD, Principal Investigator — Worldwide Clinical Trials Early Phase Services
Locations (1):
- Worldwide Clinical Trials Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No